CLINICAL TRIAL: NCT05930171
Title: Analgesic Efficacy of Combined Lumbar Erector Spinae Plane Block and Pericapsular Nerve Group Block in Patients Undergoing Hip Surgeries
Brief Title: Combined Lumbar Erector Spinae Plane Block and Pericapsular Nerve Group Block in Patients Undergoing Hip Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ibrahim Walash, Assistant Lecturer of anesthesia, intensive care and pain management, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Lumbar ESPB and PENG block
Record Dates: First submitted 2023-06-04; First posted 2023-07-05 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Lumbar Erector Spinae Plane Block; Pericapsular Nerve Group Block (PENG Block)
Keywords: Lumbar Erector Spinae Plane Block; Pericapsular Nerve Group Block; Hip Surgeries; L-ESPB; PENG block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: L-ESPB and PENG (Active Comparator): receiving after end of hip surgery (PENG) block first and (LESPB) at lumber 4 vertebrae level
  Interventions: Procedure: Ultrasound guided L-ESPB and PENG block using Bupivacaine
- Group B: conventional analgesia (Active Comparator): receiving postoperative conventional analgesia in form of acetaminophen 15 mg/kg/6hrs
  Interventions: Drug: Postoperative conventional analgesia in form of Acetaminophen

INTERVENTIONS:
Procedure: Ultrasound guided L-ESPB and PENG block using Bupivacaine — Combined Lumbar Erector Spinae Plane Block and Pericapsular Nerve Group Block in Patients Undergoing Hip Surgeries
  Other Names: Lumbar Erector Spinae Plane Block and Pericapsular Nerve Group Block
  Arms: Group A: L-ESPB and PENG
Drug: Postoperative conventional analgesia in form of Acetaminophen — Postoperative conventional analgesia in form of acetaminophen 15 mg/kg/6hrs
  Other Names: Conventional analgesia
  Arms: Group B: conventional analgesia

SUMMARY:
The investigators are going to evaluate the postoperative analgesic efficacy of combined LESPB and PENG block after hip surgeries.

DETAILED DESCRIPTION:
Hip surgeries are very common surgeries and has high postoperative pain potential. There are different ways to execute postoperative analgesia and each of them has advantages and disadvantages. As the patients submitted to this procedure are usually older and with multiple comorbidities, analgesia options with better profile of adverse effects should be preferred. Peripheral nerve block with long-acting local anesthetics is very suitable in this situation, in comparison with systemic or neuraxial opioids.

Pain control after total hip arthroplasty (THA) can be challenging because of complex innervation of the hip joint from both the lumbar and sacral nerve plexus. pain was the cause of 12% of unplanned hospital patient admissions, 60% of these patients were admitted for orthopedic concerns. The consequences of severe postoperative pain are prolonged hospital stay, increase hospital readmission, precipitation in the use of opioids with subsequent increase in postoperative nausea and vomiting, and overall low patient satisfaction. Furthermore, postoperative pain can seriously impact the physical and mental health of the patient and lead to secondary complications such as nausea, vomiting, slowed bowel movements, muscle spasms, thrombosis, cardiopulmonary complications and delayed recovery of organ functions.

The hip joint is innervated by the articular branches of multiple nerves that emerge from the lumbosacral plexus (L2-S1). The nerve supply to a specific region of the joint typically corresponds to the innervation of the muscle that crosses it :-

* The femoral nerve innervates the anterior aspect
* The obturator nerve supplies the inferior aspect
* The superior gluteal nerve supplies the superior aspect
* The nerve to the quadratus femoris innervates the posterior aspect.

Hip joint capsular innervation was found to consistently involve the femoral and obturator nerves, which supply the anterior capsule, and the nerve to the quadratus femoris, which supplies the posterior capsule.

Lumbar erector spinae plane block (LESPB) local anesthetics spread to lumbar paravertebral space and lumbar nerve roots, reaching the nerves responsible for the innervation of the hip joint lumbar plexus nerves - femoral, obturator and lateral femoral cutaneous nerves - providing analgesia for hip surgery. LESPB can be a block easier to perform than other options for hip surgery analgesia, such as posterior lumbar plexus.

(L-ESPB) is an effective analgesic technique after hip surgeries. However, an insufficient sensorial blockade of the medial part of the thigh which is innervated by the obturator nerve.

The pericapsular nerve group (PENG) block is an ultrasound-guided approach, first described by Giron-Arango et al. for the blockade of the articular branches of the femoral, obturator and accessory obturator nerves that provide sensory innervation to the anterior hip capsule. It has been successfully used as an alternative regional anaesthesia technique for the management of acute pain after hip fracture, but its applications are expanding, suggesting a potential role for analgesia after elective hip surgery.

After all the investigators hypothesize that combination of LESPB and PENG block can be more effective in pain control after hip surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 years old
* American Society of Anesthesiologists (ASA) class I to III
* Both sex
* Scheduled for hip surgery.

Exclusion Criteria:

* Refusal to participate
* Allergy to any of the study drugs
* Bleeding disorder
* Localized infection
* Neurological disease
* Renal impairment
* Psychological disorders
* Opioid dependent
* Intellectual disability (patients unable to express pain with visual analogue)
* Morbid obesity.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain intensity | at 1 hour after the block
  Postoperative pain intensity using Visual Analogue Scale (VAS) (which is over 10 centimeter scale) (where 0 indicates no pain at all , 10 indicates severe pain)
Postoperative pain intensity | at 3 hour after the block
  Postoperative pain intensity using Visual Analogue Scale (VAS) (which is over 10 centimeter scale) (where 0 indicates no pain at all , 10 indicates severe pain)
Postoperative pain intensity | at 6 hour after the block
  Postoperative pain intensity using Visual Analogue Scale (VAS) (which is over 10 centimeter scale) (where 0 indicates no pain at all , 10 indicates severe pain)
Postoperative pain intensity | at 12 hour after the block
  Postoperative pain intensity using Visual Analogue Scale (VAS) (which is over 10 centimeter scale) (where 0 indicates no pain at all , 10 indicates severe pain)
Postoperative pain intensity | at 24 hour after the block
  Postoperative pain intensity using Visual Analogue Scale (VAS) (which is over 10 centimeter scale) (where 0 indicates no pain at all , 10 indicates severe pain)

SECONDARY OUTCOMES:
Vital signs | assessed at preoperative, postoperative (0,3,6,12,24 hours), Value is averaged of total measurements
  Heart Rate
Vital signs | assessed at preoperative, postoperative (0,3,6,12,24 hours), Value is averaged of total measurements
  Arterial Blood Pressure
Vital signs | assessed at preoperative, postoperative (0,3,6,12,24 hours), Value is averaged of total measurements
  Arterial Oxygen Saturation
Time to first analgesic administration | 24 hours postoperative
  Time to first analgesic administration
Total Analgesic Requirements | 24 hours postoperative
  Total analgesic requirements in 24 hours postoperative
Patient satisfaction | 24 hours after the block
  patients will be asked to assess their satisfaction :-
  * I Very satisfied.
  * II sometimes satisfied.
  * III Neither satisfied nor dissatisfied.
  * IV Somewhat dissatisfied.
  * V Very dissatisfied.
Adverse events | 24 hours after the block
  Either hematoma, infection, postoperative nausea, vomiting orlocal anesthetic systemic toxicity
Block failure (patients still feeling pain immediately after 1 hour from block) | 1 hour after the block
  Block failure (patients still feeling pain immediately after 1 hour from block)

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia university, Menoufia, Menoufia, Egypt

REFERENCES:
- [Background] Ahiskalioglu A, Tulgar S, Celik M, Ozer Z, Alici HA, Aydin ME. Lumbar Erector Spinae Plane Block as a Main Anesthetic Method for Hip Surgery in High Risk Elderly Patients: Initial Experience with a Magnetic Resonance Imaging. Eurasian J Med. 2020 Feb;52(1):16-20. doi: 10.5152/eurasianjmed.2020.19224. PMID 32158307
- [Background] Santonastaso DP, De Chiara A, Kraus E, Bagaphou TC, Tognu A, Agnoletti V. Ultrasound guided erector spinae plane block: an alternative technique for providing analgesia after total hip arthroplasty surgery? Minerva Anestesiol. 2019 Jul;85(7):801-802. doi: 10.23736/S0375-9393.19.13459-1. Epub 2019 Mar 12. No abstract available. PMID 30871306
- [Background] Tulgar S, Kose HC, Selvi O, Senturk O, Thomas DT, Ermis MN, Ozer Z. Comparison of Ultrasound-Guided Lumbar Erector Spinae Plane Block and Transmuscular Quadratus Lumborum Block for Postoperative Analgesia in Hip and Proximal Femur Surgery: A Prospective Randomized Feasibility Study. Anesth Essays Res. 2018 Oct-Dec;12(4):825-831. doi: 10.4103/aer.AER_142_18. PMID 30662115
- [Background] Tulgar S, Selvi O, Senturk O, Ermis MN, Cubuk R, Ozer Z. Clinical experiences of ultrasound-guided lumbar erector spinae plane block for hip joint and proximal femur surgeries. J Clin Anesth. 2018 Jun;47:5-6. doi: 10.1016/j.jclinane.2018.02.014. Epub 2018 Mar 6. No abstract available. PMID 29522966
- [Background] Tulgar S, Senturk O. Ultrasound guided Erector Spinae Plane block at L-4 transverse process level provides effective postoperative analgesia for total hip arthroplasty. J Clin Anesth. 2018 Feb;44:68. doi: 10.1016/j.jclinane.2017.11.006. Epub 2017 Nov 14. No abstract available. PMID 29149734
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Del Buono R, Padua E, Pascarella G, Costa F, Tognu A, Terranova G, Greco F, Fajardo Perez M, Barbara E. Pericapsular nerve group block: an overview. Minerva Anestesiol. 2021 Apr;87(4):458-466. doi: 10.23736/S0375-9393.20.14798-9. Epub 2021 Jan 12. PMID 33432791
- [Background] Lin DY, Morrison C, Brown B, Saies AA, Pawar R, Vermeulen M, Anderson SR, Lee TS, Doornberg J, Kroon HM, Jaarsma RL. Pericapsular nerve group (PENG) block provides improved short-term analgesia compared with the femoral nerve block in hip fracture surgery: a single-center double-blinded randomized comparative trial. Reg Anesth Pain Med. 2021 May;46(5):398-403. doi: 10.1136/rapm-2020-102315. Epub 2021 Feb 26. PMID 33637625
- [Background] Del Buono R, Padua E, Pascarella G, Soare CG, Barbara E. Continuous PENG block for hip fracture: a case series. Reg Anesth Pain Med. 2020 Oct;45(10):835-838. doi: 10.1136/rapm-2020-101446. Epub 2020 Aug 12. PMID 32796133
- [Background] Roy R, Agarwal G, Pradhan C, Kuanar D. Total postoperative analgesia for hip surgeries, PENG block with LFCN block. Reg Anesth Pain Med. 2019 Mar 28:rapm-2019-100454. doi: 10.1136/rapm-2019-100454. Online ahead of print. No abstract available. PMID 30923252
- [Background] Kukreja P, Schuster B, Northern T, Sipe S, Naranje S, Kalagara H. Pericapsular Nerve Group (PENG) Block in Combination With the Quadratus Lumborum Block Analgesia for Revision Total Hip Arthroplasty: A Retrospective Case Series. Cureus. 2020 Dec 23;12(12):e12233. doi: 10.7759/cureus.12233. PMID 33500856

DOCUMENTS (2):
  • Study Protocol (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT05930171/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT05930171/SAP_001.pdf